CLINICAL TRIAL: NCT01495871
Title: Amino Acid Supplementation in Recovery From Traumatic Brain Injury
Acronym: TBIS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decided not to pursue this study.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: The Moody Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 10-276
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Amino Acids; Valine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Amino acids (Active Comparator): Amino acid supplementation for 6 weeks
  Interventions: Dietary Supplement: Amino Acids
- Placebo (Placebo Comparator): Supplementation of placebo (inert components)for 6 weeks
  Interventions: Dietary Supplement: Placebo of inert compounds
- Valine (Active Comparator): Valine supplementation for 6 weeks
  Interventions: Dietary Supplement: Valine

INTERVENTIONS:
Dietary Supplement: Amino Acids — 15 grams amino acids two times per day for 6 weeks
  Arms: Amino acids
Dietary Supplement: Placebo of inert compounds — Placebo two times per day for 6 weeks
  Arms: Placebo
Dietary Supplement: Valine — 2.5 grams valine supplementation two times a day for 6 weeks
  Arms: Valine

SUMMARY:
Traumatic brain injury (TBI) is a leading cause of death and disability in young people. It has been called the "signature wound" of the Iraq war because of its frequency among troops. TBI is associated with many chronic disabilities. Physical alterations include reduced exercise tolerance and profound muscle weakness, whereas psychological alterations include diminished sense of well-being, depression, fatigue and anxiety. Muscle and brain tissues rely upon circulating blood amino acids as precursors for metabolic functions. The investigators have shown that even one year after injury, plasma valine, an essential amino acid (EAA), was markedly reduced in patients with TBI compared to healthy controls. The investigators speculate that low plasma valine concentration contributes to chronic fatigue after TBI, since valine and tryptophan compete for the same transporter into the brain, and a low plasma valine concentration will allow more tryptophan to be transported. As a consequence, increased brain tryptophan will increase serotonin production, which may significantly contribute to the development of fatigue. Thus, the investigators will test if restoring valine concentration in persons with TBI may reduce fatigue perception and improve physical and neuropsychological function. Further, the investigators have previously shown that EAA intake has an anabolic effect in healthy young and elderly individuals. However, no data are currently available in persons recovering from TBI. Thus,the investigators will also test if EAA and/or valine can improve muscle mass in patients with TBI.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of traumatic brain injury
2. Age 18-65 years
3. Ability to sign informed consent
4. >3 months post-injury, <36 months post-injury
5. Ambulatory or require minimal to moderate assistance for safe ambulation

Exclusion Criteria:

1. Subjects with cardiac abnormalities considered exclusionary by the study physicians
2. Subjects with uncontrolled metabolic disease, including liver or renal disease
3. Subjects with cancer or recently (6 months) treated cancer other than basal cell carcinoma
4. Any subject currently on a weight-loss diet or a body mass index >34 kg/m2
5. Recent anabolic or corticosteroids use (within 3 months)
6. Dementia
7. Inability to tolerate an upright position
8. Postural reflexes prohibiting ambulation and inability to follow 2-step commands
9. Any other condition or event considered exclusionary by the PIs and covering physician

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Essential Amino Acid Concentrations | 6 weeks
  TBI patients are deficient in a number of essential amino acids (EAA) post injury and we have shown that TBI patient are deficient in valine up to 17 months post injury. We propose to assess plasma amino acid concentrations in TBI patients who are receiving EAA supplementation or valine supplementation compared to placebo patients.

SECONDARY OUTCOMES:
Functional impairments | 6 weeks
  Reduced plasma EAAs may be related to the psychological and metabolic complications associated with TBIs. We aim to assess measures of psychological and physical functionality in TBI patients receiving EAA supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Sheffield-Moore, Ph.D., Principal Investigator — The University of Texas Medical Branch, Galveston
Locations (2):
- United States (2):
  - Transitional Learning Center, Galveston, Texas
  - University of Texas Medical Branch, Galveston, Texas